CLINICAL TRIAL: NCT01922778
Title: Screening for Endometrial Abnormalities in Overweight and Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-0105
Record Dates: First submitted 2013-08-08; First posted 2013-08-14 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Endometrial Biopsy (Experimental): Recruits from the Bariatric Surgery Program will be interviewed by a study investigator prior to their bariatric surgery. If the patient consents to the procedure, then this will usually be a D&C performed in one setting at the time of her bariatric surgery under general anesthesia. In the case where a patient is diagnosed with complex atypical endometrial hyperplasia or early endometrial prior to her bariatric surgery, an IUD device can be inserted at the time of her bariatric surgery.
  For patients not undergoing bariatric surgery, an endometrial biopsy will be performed in the clinic or office setting. If the biopsy cannot be performed due to technical difficulty (cervical stenosis) or inadequate sampling, we will try again on a different day after a trial of vaginal misoprostol (Cytotec) 400 or 600 mcg per vagina the night before.
  Interventions: Procedure: Endometrial Biopsy

INTERVENTIONS:
Procedure: Endometrial Biopsy — Recruits from the Bariatric Surgery Program will be interviewed by a study investigator prior to their bariatric surgery. During the interview, the purpose of the study will be explained as well as the surgical technique used for obtaining an endometrial sample. If the patient consents to the procedure, then this will usually be a D&C performed in one setting at the time of her bariatric surgery under general anesthesia. In the case where a patient is diagnosed with complex atypical endometrial hyperplasia or early endometrial prior to her bariatric surgery, an IUD can be inserted at the time of her bariatric surgery.
  For patients not undergoing bariatric surgery, an endometrial biopsy will be performed in the clinic or office setting using an endometrial suction catheter.

SUMMARY:
The purpose of this study is to develop an endometrial biopsy screening program for endometrial cancer and its precursor lesions in overweight and obese women.

There is a BMI threshold at and above which optimal screening parameters exist for identifying endometrial cancer and its precursor lesions in overweight and/or obese women. Prevention, diagnosis and treatment of endometrial cancer and its precursor lesions in overweight and/or obese women offers substantial health benefits.

ELIGIBILITY:
INCLUSION CRITERIA:

* Have BMI ≥25.
* Be patients of the St. Luke's and Roosevelt Gynecology Clinics and Faculty Practices OR be receiving bariatric surgery.
* Complete a full medical history, a detailed menstrual and/or postmenopausal bleeding history, and endometrial biopsy.
* Have a negative pregnancy test, if of childbearing age.
* Be at least 18 years of age.
* Have signed a written Informed Consent Document.
* Be willing and able to comply with the study requirements.

EXCLUSION CRITERIA:

* Have a BMI <25.
* Have a prior hysterectomy.
* Be pregnant or have a positive pregnancy test
* Have untreated vaginal, cervical, or adnexal infection.
* Recent treatment of STD

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2013-09; Primary Completion 2016-03-31 (Actual); Study Completion 2016-03-31 (Actual)

PRIMARY OUTCOMES:
A BMI cut-point will be identified at and above which an endometrial biopsy yields optimal sensitivity, specificity, positive predictive value, and negative predictive value to screen for endometrial cancer and abnormal pathologies | up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Anderson, MD, Principal Investigator — Mount Sinai Roosevelt
Locations (1):
- Mount Sinai Roosevelt, New York, New York, United States